CLINICAL TRIAL: NCT03687151
Title: Population-based Cancer Observatory of the French Region Sud-Provence-Alpes-Côte d'Azur Recruiting Incident Cases of Cancer Since 2005
Brief Title: Population-based Cancer Observatory
Acronym: cancer observ
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-DSP-04
Record Dates: First submitted 2018-09-20; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with a diagnosis of invasive or in situ cancer: patients with a diagnosis of invasive or in situ cancer living in the French Region Sud-Provence-Alpes-Côte d'Azur since 2005
  Interventions: Other: non intervention / observationnal

INTERVENTIONS:
Other: non intervention / observationnal — non intervention / observationnal

SUMMARY:
Cancer is the leading cause of death in Western countries. In France cancer control plans (National screening programmes) and recommendations for the management of cancer patients (multidisciplinary team meetings), have been implemented. Evaluating the effectiveness of these policies aiming for improved prevention and management is essential. However to conduct such an evaluation, a baseline reference requiring ongoing, reliable and complete data collection is necessary and can be used for epidemiological research.

There is no cancer registry in the French Region Sud-Provence-Alpes-Côte d'Azur. In view of this situation, the regional Health Agency appointed the public health department of the Nice Côte d'Azur University and the Centre for computerized pathology data collection (CRISAP-PACA) to develop a Cancer Observatory. Since 2005, the public health department collects data concerning invasive and in situ cancers from all the histopathology labs in the French Region Sud-Provence-Alpes-Côte d'Azur, gathered in the CRISAP-PACA, and transmits incidence cancer rates to the regional Health Agency. In 2007, a quality control procedure, comparing a random sample of data collected by the Cancer Observatory with pathology lab reports, confirmed the validity of the collected data with fewer than 3% in disagreement with the report's conclusions. In 2008, the estimated completeness of cancer records collected from histopathology laboratories was higher than 90% for new cases of breast and colorectal cancer within the age range concerned by the screening programme. Since 2012, public and private hospitals treating cancer patients as well as the regional cancer network ONCOPACA, coordinating multiple team meetings, have been contacted to transmit to the public health department cases of cancer without histological diagnosis. In addition, patients with cancer have been geolocated to study the influence of environmental exposures on the occurrence of cancers (patients living near of waste incinerator, highways).

ELIGIBILITY:
Inclusion Criteria:

* All subjects with a diagnosis of invasive or in situ cancer living in the French Region Sud-Provence-Alpes-Côte d'Azur.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with cancer
Sampling Method: Non-Probability Sample
Dates: Start 2005-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
number of each cancer of the French Region Sud-Provence-Alpes-Côte d'Azur | 50 years
  each cancer is definite by :number of Date of diagnosis, Tumor location, Histology, ADICAP codes, CIM-O codes, Age, Gender and Geolocation.
  number of classification of cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No